CLINICAL TRIAL: NCT00882622
Title: Effect of Remote Ischemic Preconditioning on Cardiac Function After Cardiac Surgery
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Endpoints were investigated in parallel in NCT00877305
Sponsor: Patrick Meybohm (Other)
Collaborators: Goethe University (Other)
Responsible Party: Sponsor-Investigator, Patrick Meybohm, PD Dr., University Hospital Schleswig-Holstein
Organization: University Hospital Schleswig-Holstein (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A165/08_2
Record Dates: First submitted 2009-04-14; First posted 2009-04-16 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Atrial Fibrillation; Ventricular Arrythmias; Myocardial Injury; Cardiac Function
Keywords: Ischemic Preconditioning; Cardiac Surgery
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RIPC (Active Comparator)
  Interventions: Procedure: Remote Ischemic Preconditioning
- CONTROL (Sham Comparator)
  Interventions: Procedure: Control/sham procedure

INTERVENTIONS:
Procedure: Remote Ischemic Preconditioning — RIPC will be induced during anesthesia by four 5-min cycles of upper limb ischemia and 5-min reperfusion using a blood-pressure cuff inflated to a pressure 15 mm Hg greater than the systolic arterial pressure measured via the arterial line.
  Arms: RIPC
Procedure: Control/sham procedure — Sham placement of the blood pressure cuff around the upper limb without inflation.
  Arms: CONTROL

SUMMARY:
The purpose of this study is to evaluate the effects of Remote Ischemic Preconditioning on cardiac function in patients undergoing cardiac surgery compared to control intervention.

DETAILED DESCRIPTION:
In detail, we will focus on new onset of atrial fibrillation, ventricular arrhythmias, myocardial injury, and cardiac function. Furthermore, we aim to investigate underlying pathways of RIPC in modifying the perioperative stress response.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing heart surgery on cardiopulmonary bypass

Exclusion Criteria:

* Emergency cases
* Myocardial infarction up to 7 days prior to enrollment
* Ejection fraction less than 30%
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-02; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
New onset of atrial fibrillation | Within 30 days after surgery

SECONDARY OUTCOMES:
Ventricular arrhythmias, myocardial injury, cardiac function. Underlying pathways of Remote Ischemic Preconditioning in modifying the perioperative stress response. | Within 24 hours after surgery

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University Hospital, Frankfurt am Main
  - University Hospital Schleswig-Holstein, Kiel